CLINICAL TRIAL: NCT00072384
Title: A Single Arm Trial of Systemic And Subtenon Chemotherapy For Groups C And D Intraocular Retinoblastoma
Brief Title: Systemic Chemotherapy and Subtenon Carboplatin, and Local Ophthalmic Therapy in Children With Intraocular Retinoblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARET0231; NCI-2009-00420 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000339627 (Other: Clinical Trials.gov); COG-ARET0231 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Intraocular Retinoblastoma
MeSH Terms: interventions — Vincristine; Cryosurgery; Laser Therapy; Carboplatin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, surgery) (Experimental): Patients receive liposomal vincristine sulfate IV over 1 minute on day 1 and carboplatin IV over 1 hour and etoposide IV over 1 hour on days 1 and 2. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 3 and continuing until blood counts recover. Patients receive subtenon carboplatin to each group C or D eye on day 0 or 1prior of courses 2-4 only. Treatment repeats every 28 days for 6 courses in the absence of occurrence of extraocular retinoblastoma or a second malignancy. Beginning with course 3 of systemic chemotherapy, patients undergo local ophthalmic therapy comprising local laser surgery and/or cryosurgery on day 1.
  Interventions: Drug: liposomal vincristine sulfate; Procedure: cryosurgery; Procedure: laser surgery; Drug: carboplatin; Drug: etoposide; Biological: filgrastim

INTERVENTIONS:
Drug: liposomal vincristine sulfate — Given IV
  Other Names: liposomal vincristine; Marqibo; vincristine liposomal; vincristine sulfate liposome injection
Procedure: cryosurgery — Application of extreme cold to destroy abnormal or diseased tissue.
  Other Names: cryoablation; cryosurgical ablation
Procedure: laser surgery — Surgery using a laser (instead of a scalpel) to cut tissue
  Other Names: conventional laser therapy; laser therapy, conventional; surgery, laser
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Biological: filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen

SUMMARY:
Phase III trial to determine the effectiveness of combining systemic chemotherapy and subtenon carboplatin with ophthalmic therapy in treating children who have intraocular retinoblastoma. Drugs used in chemotherapy, such as vincristine, carboplatin, and etoposide, work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether systemic chemotherapy and subtenon (under the conjunctiva of the eye) carboplatin combined with ophthalmic therapy is effective in treating intraocular (within the eyeball) retinoblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the event-free survival at 12 months of pediatric patients' eyes with group D intraocular retinoblastoma treated with systemic chemotherapy comprising vincristine, carboplatin, and etoposide, subtenon carboplatin, and local ophthalmic therapy. (Event defined for each eye individually as needed for nonprotocol therapy including nonprotocol chemotherapy, enucleation or any external-beam radiation)

SECONDARY OBJECTIVES:

I. Determine the event-free survival at 12 months of pediatric patients' eyes with group C retinoblastoma treated with systemic chemotherapy comprising carboplatin, etoposide, vincristine, subtenon carboplatin, and local ophthalmic therapy.

II. Determine the acute and long-term toxic effects of these regimens in these patients, including visual outcome and incidence of secondary malignancies.

III. Determine the patterns of failure in patients treated with these regimens, in terms of vitreous vs retinal vs both as sites of recurrence.

IV. Determine predictors of failure including findings at the on study examination under anesthesia and response status after six courses of chemotherapy.

V. Determine the percentage of group C and D eyes separately that can be preserved without enucleation after failing protocol therapy.

OUTLINE: This is a multicenter study.

Patients receive vincristine IV over 1 minute on day 1 and carboplatin IV over 1 hour and etoposide IV over 1 hour on days 1 and 2. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 3 and continuing until blood counts recover. Patients receive subtenon carboplatin to each group C or D eye on day 0 or 1 prior of courses 2-4 only. Treatment repeats every 28 days for 6 courses in the absence of occurrence of extraocular retinoblastoma or a second malignancy. Beginning with course 3 of systemic chemotherapy, patients undergo local ophthalmic therapy comprising local laser and/or cryotherapy on day 1.

Patients are followed with ophthalmology exams every 4-12 weeks until 3 years of age, every 6 months until 5 years of age, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral retinoblastoma with at least 1 eye group C or D intraocular retinoblastoma by ophthalmologic examination, defined by the International Classification System for Intraocular Retinoblastoma as the following:

  * Group C: Discrete localized disease with minimal subretinal and/or vitreous seeding

    * Subretinal fluid, without prior or concurrent seeding, involving ≤ one quarter of the retina
    * Local fine vitreous seeding may be present close to discrete tumor
    * Local subretinal seeding < 3 mm from tumor
  * Group D: Diffuse disease with significant vitreous and/or subretinal seeding

    * Tumor(s) may be massive or diffuse
    * Subretinal fluid, without prior or concurrent seeding, involving up to total retinal detachment
    * Diffuse or massive vitreous disease may include "greasy" seeds or avascular tumor masses
    * Diffuse subretinal seeding may include subretinal plaques or tumor nodules
* Prior enucleation of 1 eye allowed provided the remaining eye is group C or D
* No tumor present on histologic examination at the cut end of the optic nerve on any eye enucleated prior to study entry

  * Evidence of choroidal and/or optic nerve invasion past the lumina cribrosa is allowed
* No extraocular retinoblastoma clinically or by MRI of brain and orbits with and without gadolinium or CT scan with and without contrast of brain and orbits
* No evidence of systemic metastases by bone marrow, lumbar puncture, bone scan, and/or any other additional test
* Performance status - Karnofsky 50-100% (over 16 years of age)
* Performance status - Lansky 50-100% (16 and under)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* AST and ALT < 2.5 times ULN for age
* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male])
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min/1.73m^2
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test in postmenarchal females
* No prior chemotherapy
* No other concurrent chemotherapy
* No prior radiotherapy
* No other concurrent radiotherapy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2007-04-16 (Actual); Primary Completion 2013-02-01 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rima Jubran, Principal Investigator — Children's Oncology Group
Locations (11):
- United States (11):
  - Children's Oncology Group, Arcadia, California
  - Southern California Permanente Medical Group, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Surgery)
Started | 30
Completed | 21
Not Completed | 9
Not completed — Physician Decision | 1
Not completed — Ineligible | 8

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Surgery)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: months] | 7.5 [1 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 12
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Group D Eyes - Treatment Failure Within One Year
Description: Each Group D eye will be classified as experiencing failure within one year after start of treatment: yes or no. The method of Rosner et al. (Biometrics v. 38, 105-114, 1982) will be used to model possible dependence between eyes from the same patient. The point estimate of the probability of treatment failure is reported as the "Mean" measure type.
Time Frame: One year
Population: Twenty eligible patients had at least one Group D eye to contribute to the analysis. A total of 25 Group D eyes were available for analysis.
Measure: Mean (Standard Deviation); unit: Probability of treatment failure
Units Other Than Participants: Eyes
Arm/Group | Treatment (Chemotherapy, Surgery)
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 25
Probability of treatment failure | 0.52 (0.102299)

2. Primary Outcome: Group C Eyes - Treatment Failure Within One Year
Description: Each Group C eye will be classified as experiencing failure within one year after start of treatment: yes or no. The method of Rosner et al. (Biometrics v. 38, 105-114, 1982) will be used to model possible dependence between eyes from the same patient. The point estimate of the probability of treatment failure is reported as the "Mean" measure type.
Time Frame: One year
Population: Four eligible patients had at least one Group C eye to contribute to the analysis
Measure: Mean (Standard Deviation); unit: Probability of treatment failure
Units Other Than Participants: Eyes
Arm/Group | Treatment (Chemotherapy, Surgery)
Number analyzed (Participants) | 4
Number analyzed (Eyes) | 4
Probability of treatment failure | 0.25 (0.217)

3. Secondary Outcome: Event-free Survival (EFS)
Description: Proportion of patients event free at 1 year following enrollment. Event free survival time is computed as the time to study entry until disease relapse/progression, secondary malignancy, or death.
Time Frame: One year after study enrollment
Population: 22 eligible patients were considered for this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage probability
Arm/Group | Treatment (Chemotherapy, Surgery)
Number analyzed (Participants) | 22
Percentage probability | 45.45 [24.44 to 64.33]

4. Secondary Outcome: Toxicity Associated With Chemotherapy
Description: The number of patients that experience CTC Version 4 grade 3 or higher toxicities of any kind.
Time Frame: From date of enrollment until termination of protocol therapy assessed up to 72 weeks
Population: 22 eligible patients were evaluable for the occurrence of grade 3 or higher toxicity of any kind.
Measure: Number; unit: Patients
Arm/Group | Treatment (Chemotherapy, Surgery)
Number analyzed (Participants) | 22
Patients | 10

5. Secondary Outcome: Patterns of Failure for Group C and Group D in Terms of Vitreous vs Patterns of Failure for Group C and Group D in Terms of Vitreous vs Retinal vs Both as Sites of Recurrence
Description: Sites of disease recurrence for Group C and Group D eyes where treatment failure was detected
Time Frame: From the date of enrollment assessed up to 36 months
Population: 1 patient had at least one Group C eye and 11 patients had at least one Group D eye that experienced treatment failure. There were a total of 13 Group D eyes that experienced treatment failure.
Measure: Number; unit: Eyes
Groups:
- Group C Eyes: Group C: Discrete localized disease with minimal subretinal and/or vitreous seeding
  * Subretinal fluid, without prior or concurrent seeding, involving ≤ one quarter of the retina
  * Local fine vitreous seeding may be present close to discrete tumor
  * Local subretinal seeding < 3 mm from tumor
- Group D Eyes: Group D: Diffuse disease with significant vitreous and/or subretinal seeding
  * Tumor(s) may be massive or diffuse
  * Subretinal fluid, without prior or concurrent seeding, involving up to total retinal detachment
  * Diffuse or massive vitreous disease may include "greasy" seeds or avascular tumor masses
  * Diffuse subretinal seeding may include subretinal plaques or tumor nodules
Arm/Group | Group C Eyes | Group D Eyes
Number analyzed (Participants) | 1 | 11
Eyes
  Retinal seeding and vitreal seeding | 0 | 1
  Retinal seeding but no vitreal seeding | 1 | 7
  Vitreal seeding but no retinal seeding | 0 | 1
  Neither retinal seeding nor vitreal seeding | 0 | 4

6. Secondary Outcome: Patterns of Treatment Failure vs. no Treatment Failure for Group C Eyes and Group D Eyes According to Initial Sites of Involvement
Description: The association between the probability of experiencing treatment failure vs. no failure in a C eye and the presence of subretinal seeding (SRS), subretinal fluid (SRF), or vitreal seeding (VS) at the on study ophthalmological examination under anesthesia. The association between the probability of experiencing treatment failure vs. no failure in a D eye and the presence of subretinal seeding (SRS), subretinal fluid (SRF), or vitreal seeding (VS) at the on study ophthalmological examination under anesthesia.
Time Frame: From the date of enrollment assessed up to 12 months
Population: According to the initial sites of involvement, 4 patients were analyzed in Group C eyes and 20 patients were analyzed for Group D eyes
Measure: Number; unit: Eyes
Arm/Group | Group C Eyes | Group D Eyes
Number analyzed (Participants) | 4 | 20
Eyes
  Treatment failure- SRS, SRF, VS | 0 | 3
  Treatment failure- SRS; no SRF; no VS | 0 | 0
  Treatment failure- SRS and SRF; no VS | 0 | 3
  Treatment failure- SRS and VS; no SRF | 0 | 0
  Treatment failure- SRF; no SRS; no VS | 1 | 2
  Treatment failure- SRF and VS; no SRS | 0 | 3
  Treatment failure- VS; no SRS; no SRF | 0 | 2
  Treatment failure- No SRS; no VS; no SRF | 0 | 0
  No treatment failure- SRS, SRF, VS | 0 | 2
  No treatment failure- SRS; no SRF; no VS | 0 | 1
  No treatment failure- SRS and SRF; no VS | 0 | 2
  No treatment failure- SRS and VS; no SRF | 0 | 2
  No treatment failure- SRF; no SRS; no VS | 1 | 2
  No treatment failure- SRF and VS; no SRS | 0 | 0
  No treatment failure- VS; no SRS; no SRF | 1 | 2
  No treatment failure- No SRS; no VS; no SRF | 1 | 1

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Note that while the participant flow demonstrates that 21 completed all cycles of therapy, one additional patient completed fewer than 6 cycles of therapy. The AE profiles are calculated on a per-person basis for the time during which the patient was on therapy.
Arm/Group | Treatment (Chemotherapy, Surgery)
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 18/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, Surgery) (N=22)
Anorectal infection (Infections and infestations) | 1
Bladder infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Eye infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.